CLINICAL TRIAL: NCT04295434
Title: Study of the European Society of Hypertension on Blood Pressure Control in ESH Excellence Centres
Brief Title: Blood Pressure Control in ESH Excellence Centres
Acronym: BP-CON
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Clinical Hospital Centre Zagreb (Other)
Collaborators: European Society of Hypertension (Other)
Responsible Party: Principal Investigator, Prof. Bojan Jelaković, Professor, Clinical Hospital Centre Zagreb
Other Study IDs: BP-CON-ESH
Record Dates: First submitted 2020-02-26; First posted 2020-03-04 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Blood Pressure; Lifestyle Risk Reduction; White Coat Hypertension
Keywords: Blood pressure; Hypertension; Control; European; Excellence centres
MeSH Terms: conditions — Risk Reduction Behavior; White Coat Hypertension; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the BP-CON-ESH study we are going to include and analyze treated hypertensive patients seen consecutively by the ESH Excellence Centres. Blood pressure will be measured as usually done in the office, but care will be adopted to make measurements highly standardized in all Centres. The primary goals will be to determine the global, regional and country rates of hypertension control in Europe. Other goals will be to identify global and regional factors associated with blood pressure control in different European regions. The results obtained in the BP-CON-ESH project will be used to refine treatment strategies for improvement of blood pressure control and will serve as a basis for assessing future changes and trends in Europe.

DETAILED DESCRIPTION:
The most important task of the European Society of Hypertension is to improve blood pressure treatment and increase blood pressure control, thus decreasing cardiovascular risk, premature cardiovascular and renal morbidity and mortality, with in addition a reduction of health-care costs. More than a decade ago, the European Society of Hypertension established a network of Excellence Centres. Those centres are leading institutions for the diagnosis and treatment of hypertension and thus are front runners of good clinical practice in hypertension management in their countries. An important task of the Excellence Centres is also to be active in research, particularly in projects conducted by the European Society of Hypertension. The ongoing BP-CON-ESH project on the rate of blood pressure control in hypertensive patients addresses the most elementary,but at the same timethe most important aspect in hypertension management, because the observed low rates of blood pressure control is the reason why hypertension is still today the leading cause of death worldwide.

In the BP-CON-ESH study we are going to include and analyze treated hypertensive patients seen consecutively by the ESH Excellence Centres. Blood pressure will be measured as usually done in the office, but care will be adopted to make measurements highly standardized in all Centres.

The primary goals will be to determine the global, regional and country rates of hypertension control in Europe. Other goals will be to identify global and regional factors associated with blood pressure control in different European regions. It is well known that the overall control of hypertension in Europe is still insufficient. However, the problem is not the same across Europe. Differences in healthcare systems exist among European countries, and in some countries government healthcare system only partially reimburse costs of antihypertensive therapy. There are also differences in gross national product, educational levels, salt consumption, prevalence of obesity and other aspects. These could cause dissimilarities in hypertension prevalence, achieved blood pressure control and cardiovascular mortality among European regions.

The results obtained in the BP-CON-ESH project will be used to refine treatment strategies for improvement of blood pressure control and will serve as a basis for assessing future changes and trends in Europe.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent

Exclusion Criteria:

* Pregnancy and breastfeeding
* Terminal malignancy, reduced life expectancy (<6 months)
* Amputated limb
* Dementia
* Patients living in a nursing home
* Unsigned informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hypertension that are under supervision of excellence centres participating in the study.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Blood pressure control | Through study completion, an average of 1 year
  Difference in blood pressure values between ESH Excellence Centres

CONTACTS AND LOCATIONS:
Overall Officials: Bojan Jelaković, MD, PhD, Principal Investigator — Clinical Hospital Centre Zagreb
Locations (46):
- Center of Preventive Cardiology, Yerevan, Yerevan, Armenia
- Klinikum Wels-Grieskirchen, Wels, Austria
- Belgium (3):
  - Erasmus Hospital, Brussels
  - CHU de Liège, Liège
  - Ambroise Paré University Hospital, Mons
- University Hospital "St. Anna", Sofia, Bulgaria
- University hospital centre Zagreb, Zagreb, City of Zagreb, Croatia
- Czechia (3):
  - Charles University Medical School and University Hospital, Pilsen
  - Center for Hypertension, Charles University, Prague, Prague
  - Institute for Clinical and Experimental Medicine (IKEM) and Thomayer Hospital, Prague, Prague
- Tallinn Hypertension Excellence Centre, Tallinn, Estonia
- Germany (5):
  - Hypertension Center Berlin Charité, Berlin
  - Hypertoniezentrum Bonn, Bonn
  - Medizinische Hochschule Hannover, Hanover
  - Universitätskliniken des Saarlandes, Homburg
  - Hypertension Center Munich, Munich
- Greece (10):
  - Hypertension and Cardiovascular Prevention Clinic, 3rd Department of Medicine, Evangelismos Hospital, Athens
  - Hypertension Clinic, University Hospital Laiko, Athens
  - University of Athens, Hippokration Hospital, Athens
  - Hypertension Clinic, Department of Cardiology, KAT General Hospital, Athens
  - Hypertension Clinic, Cardiology Department, Asklepeion Hospital, Athens
  - University Hospital of Heraklion, Heraklion
  - Hypertension Center, Department of Nephrology, University Hospital of Ioannina, Ioannina
  - Hypertension Outpatient Clinic, 1st Propedeutic Dept. of Internal Medicine, AHEPA Hospital, Thessaloniki
  - Hypertension Center, Department of Nephrology, Hippokration Hospital, Aristotle University of Thessaloniki, Thessaloniki
  - Aristotle University of Thessaloniki, Papageorgiou General Hospital, Thessaloniki
- Assuta Ashdod University Hospital, Ashdod, Israel
- Italy (5):
  - Centre of Prevention and Treatment of Arterial Hypertension and Cardiovascular Risk Factors, Brescia
  - S. Luca Hospital, Istituto Auxologico Italiano, Milan
  - Ospedale Niguarda, Dip. De Gasperis e Università di Milano Bicocca, Milan
  - Napoli Hypertension Excellence Centre, Federico II Clinic Research Center for Hypertension and Related Conditions, Napoli
  - Excellence Centre of Hypertension, Department of Medical Sciences, University of Torino, Torino
- American University Center, Hypertension/Vascular Medicine Division (Associated Centre), Beirut, Lebanon
- Kaunas Hypertension Excellence Centre, Kaunas, Lithuania
- Netherlands (2):
  - University Hospital Maastricht, Maastricht
  - Radboud University of Nijmegen Medical Center, Nijmegen
- Department of Internal Medicine, Hypertension and Vascular Diseases, Warsaw Medical University, Warsaw, Poland
- Centro Hospitalar do Alto Ave, Minho University, Guimarães, Portugal
- Department of Cardiology and Internal Medicine, Emergency Clinical Hospital of Bucharest, Bucharest, Romania
- Centre for Hypertension of the Clinical Centre of Serbia, Belgrade, Serbia
- Spain (2):
  - Hipertensión Clinic, Internal Medicine, Hospital Clinico, University of Barcelona, Barcelona
  - Hypertension Clinic, Nephrology Department, Reina Sofia University Hospital, Córdoba
- Danderyd University Hospital, Stockholm, Sweden
- National Scientific Center "The M.D. Strazhesko Institute of Cardiology", Kyiv, Ukraine
- United Kingdom (2):
  - St. Bartholomew's Royal London School of Medicine & Dentistry, London
  - The Pearl-Rose Clinic (Hypertension & Cardiovascular Risk), Hammersmith Hospital,, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: ESH website with relevant informations on BP CON study — https://www.eshonline.org/communities/excellence-centres/blood-pressure-control-in-esh-excellence-centres-bp-con-esh/